CLINICAL TRIAL: NCT04174196
Title: A Pilot Study Evaluating Lenalidomide and CC-486 in Combination With Radiotherapy For Patients With Plasmacytoma (LENAZART Study)
Brief Title: A Study of Lenalidomide and CC-486 With Radiation Therapy in Patients With Plasmacytoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-284
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Plasmacytoma; Plasmacytoma of Bone; Multiple Myeloma
Keywords: CC-486; Plasmacytoma; lenalidomide; Plasmacytoma of Bone; Memorial Sloan Kettering Cancer Center; 19-284; multiple myeloma with plasmacytomas; multiple myeloma
MeSH Terms: conditions — Plasmacytoma; Multiple Myeloma | interventions — cc-486; Lenalidomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Plasmacytoma (Experimental): Participants will have solitary bone plasmacytoma with minimal marrow involvement and participants with relapsed multiple myeloma with plasmacytomas
  Interventions: Drug: CC-486; Drug: Lenalidomide; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: CC-486 — Participants will be treated with CC-486 and lenalidomide for 6 cycles
Drug: Lenalidomide — Participants will be treated with CC-486 and lenalidomide for 6 cycles
Radiation: Radiation Therapy — Radiation therapy will be initiated to the plasmacytoma after cycle 2

SUMMARY:
The purpose of this study is to investigate if the combination of CC-486 with lenalidomide and radiation therapy is a safe and effective treatment for plasmacytoma.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1: Must meet all the following 3 criteria:

* Histologically confirmed newly diagnosed or recurrent solitary plasmacytoma/lytic lesion (recurrent solitary plasmacytomas will be considered based on treating physician discretion for cases where they clinically plan to treat with RT alone) - Minimal marrow involvement (Detectable clonal bone marrow plasma cells by multicolor flow cytometry and </= 10% clonal plasma cells in a bone marrow biopsy by immunohistochemistry, morphology, or flow cytometry)
* Secretory M protein < 3 g/dL

Cohort 2: Must meet all the following criteria:

* Relapsed multiple myeloma with plasmacytomas/lytic lesion appropriate for RT on imaging
* Relapsed (reappearance of M-spike/serum FLC) or progressive myeloma defined by a 25% increase from nadir in M-spike or involved serum FLB on 2 separate measurements; or with bone marrow involvement by clonal plasma cells detectable by IHC or flow cytometry.
* Any prior number of therapies is permitted, including prior radiation therapy
* Allogeneic transplant patients are permitted

All Cohorts:

* Age >/= 18 years
* Surgical resection of plasmacytoma or stabilization surgery is permitted if necessary based on physician judgement
* ECOG performance status of 0-1
* Anticipated lifespan greater than 3 months
* Able and willing to give valid written informed consent
* Creatinine clearance >/=30ml/min by Cockroft-Gault method. See section below, "Dosing Regimen", regarding lenalidomide dose adjustment for calculated creatinine clearance >/= 30ml/min and <60ml/min
* Serum bilirubin levels </= 1.5 times the upper limit of the normal range for the laboratory (ULN). Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis of Gilbert's syndrome
* AST (SGOT) and ALT (SGPT) </= 2.5 x ULN
* Women of childbearing potential should be advised to avoid becoming pregnant and must adhere to the scheduled pregnancy testing a required in the Revlimid REMS program. They must be agreeable to use acceptable methods of birth control throughout the study and for at least 6 months after the last dose:

Recommendation is for 2 effective contraceptive methods during the study and for at least 6 months after the last dose. Adequate forms of contraception are double-barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral, depo provera, or injectable contraceptive, intrauterine devices, and tubal ligation.

* Agree to abstain from breastfeeding during study participation and for at least 90 days after the last dose of investigational product (IP). Men should be advised to not father a child while receiving treatment with azacitidine. Male patients with female partners who are of childbearing potential: Recommendation is for the patient and partner use at least 2 effective contraceptive methods, as described above, during the study and for 3 months following the last dose of study drug.

Refrain from semen or sperm donation while taking IP and for at least 90 days after the last dose of IP.

* Willing to be registered into the mandatory Revlimid REMS program, and be willing and able to comply with the requirements of the REMS program.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use physician's choice of anticoagulation).
* Able to swallow oral medication
* Hematologic criteria: Hemoglobin >/= 9 g/dL, platelets >/= 50,000 and ANC >/= 1

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking azacitidine).
* Uncontrolled systemic fungal, bacterial or viral infection (defined as ongoing signs/symptoms related the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment)
* History of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), celiac disease (ie, sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the study drug and/or predispose the subject to an increased risk of gastrointestinal toxicity
* Abnormal coagulation parameters without any known etiology (PTT > 45 seconds, and/or INR > 1.5). Patients currently on therapeutic anti-coagulation treatment are exempt from these parameters.
* Significant active cardiac disease within the previous 6 months including:

NYHA class 4 CHF Unstable angina Myocardial infarction

* known or suspected hypersensitivity to azacitidine or mannitol
* Known hypersensitivity to thalidomide or lenalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) as determined by a positive Polymerase Chain Reaction (PCR) will be excluded. Patients who are seropositive because of HBV vaccine are eligible. Seropositive status-antibody positive patients with negative PCR on two occasions will be eligible
* Concurrent systemic chemotherapy with drugs other than CC-486 and lenalidomide.
* Patients on tacrolimus therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2026-11-19 (Estimated); Study Completion 2026-11-19 (Estimated)

PRIMARY OUTCOMES:
Measure Complete Response | At the end of Cycle 6 (each cycle is 28 days)
  Stringent complete response (sCR) will be computed by 2016 IMWG Criteria in addition to identifying no new lesions on PET at the end of 6 cycles of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Urvi Shah, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org